CLINICAL TRIAL: NCT06188117
Title: The Effect of Digital Game Addiction Awareness Training Given to Parents of Secondary School Students on the Awareness Level of Parents
Brief Title: Efficacy of Digital Game Addiction Awareness Training for Parent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/16-02
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Game Addiction, Video
Keywords: digital game addiction; school; parent
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The 'Digital Game Addiction Awareness Training' program will be implemented in 2 sessions in 1 day for a total of 2 hours.
  Interventions: Other: 'Digital Game Addiction Awareness Training'
- Control Group (No Intervention): The digital Game Addiction Awareness Training program will not be applied to parents in the control group.

INTERVENTIONS:
Other: 'Digital Game Addiction Awareness Training' — Experimental Group The 'Digital Game Addiction Awareness Training' program will be implemented in 2 sessions in 1 day for a total of 2 hours.
  The training program will be implemented in line with the headings 'Digital Game Addiction Definition, Diagnostic Criteria, Frequency, Symptoms, Physical, Psychological and Social Problems Caused by Excessive Digital Game Playing, Recommendations for Parents to Prevent Digital Game Addiction'.
  Arms: Experimental Group

SUMMARY:
The study will be conducted with the randomized controlled experimental method. The purpose of this research is to determine the effect of digital game addiction awareness training given to parents of 6th-grade secondary school students on their parents' awareness levels of digital game addiction. Parents will be randomly assigned to groups by lottery method. After the randomization parents of students in the intervention group will be given 'Digital Game Addiction Awareness Training'. The digital game addiction awareness level of all parents will be determined with the 'Digital Game Addiction Awareness Scale' before and 3 months after the training. Parents in the control group will not be educated. The digital game addiction awareness level of the parents in the control group will be determined with the 'Digital Game Addiction Awareness Scale' when they are included in the research and 3 months later.

DETAILED DESCRIPTION:
The use of technological devices such as computers, tablets and smartphones is increasing day by day all over the world. With the widespread use of these high-tech devices and the internet in the last 20 years, digital games have become popular as a leisure activity, especially among children and adolescents. Although digital games provide cognitive, social and emotional benefits such as improving hand-eye coordination, three-dimensional thinking, coping with stress, increasing decision-making speed and facilitating learning, excessive digital gaming can lead to psychosocial and medical problems. One of the most important problems that may develop as a result of uncontrolled use of online and offline games is digital game addiction.

Considering the addiction of digital games, it is very important to raise awareness and awareness of both children and their parents in order to protect children from the risks of digital games and to ensure that they play the games they play in a controlled manner. One of the important methods of raising awareness is to provide training to individuals on the subject for which awareness is desired. In this regard, this research was planned to examine the effect of digital game addiction awareness training on creating and increasing awareness of digital game addiction in the parents of secondary school students.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 43,
* No auditory, visual, or mental problems that would affect communication
* Speaking and understanding Turkish at native level

Exclusion Criteria:

* Being younger than 18 years old and older than 43 years old,
* Having auditory, visual, or mental problems that would affect communication
* Not speaking and understanding Turkish at native level

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Digital Game Addiction Awareness Scale | Baseline and 3 months after the Digital Game Addiction Awareness Training.
  Parents' digital game addiction awareness levels will be evaluated with the 'Digital Game Addiction Awareness Scale'. The scale is used to determine the awareness levels of individuals between the ages of 18-43 regarding digital game addiction. The scale, which consists of a total of 12 items, has two sub-dimensions: 'Internal Awareness' and 'External Awareness'. The items of the 5-point Likert type scale are rated as "1-strongly disagree", "2-disagree", "3-undecided", "4-agree" and "5-strongly agree". The scores that can be obtained from the scale vary between 12 and 60. A total scale score of the participants between 12 and 28 indicates a low level of awareness, a score between 29 and 44 indicates a moderate level of awareness, and a score between 45 and 60 indicates a high level of awareness of digital game addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Ekici, PhD, Principal Investigator — Maltepe University; Zeynep Aközlü, MSc, Principal Investigator — Maltepe University
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)